CLINICAL TRIAL: NCT04270513
Title: Flying Intervention Team for Endovascular Treatment of Acute Ischemic Stroke in Rural Areas
Acronym: FIT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Munich Municipal Hospital (Other)
Collaborators: Technical University of Munich (Other); University of Regensburg (Other)
Responsible Party: Sponsor
Other Study IDs: FIT
Record Dates: First submitted 2018-04-13; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Brain Infarction
Keywords: endovascular treatment; stroke; large vessel occlusion; telemedicine; helicopter; thrombectomy; mobile interventionalist; flying intervention team
MeSH Terms: conditions — Brain Infarction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EVT by Flying Intervention Team in primary stroke center: Patients with ischemic stroke and large vessel occlusion admitted to a primary stroke center, for whom a Flying Intervention Team is flown to the primary stroke center in order to perform endovascular treatment.
  Interventions: Other: Endovascular treatment by Flying Intervention Team
- EVT after secondary transfer to comprehensive stroke center: Patients with ischemic stroke and large vessel occlusion admitted to a primary stroke center, who are transferred to a comprehensive stroke center for endovascular treatment.

INTERVENTIONS:
Other: Endovascular treatment by Flying Intervention Team — After telemedicine-assisted decision for endovascular treatment, the Flying Intervention Team is transferred via helicopter to the primary stroke center and performs endovascular treatment in the local angiography suite.
  Groups: EVT by Flying Intervention Team in primary stroke center

SUMMARY:
The aim of this study is to compare time delay and safety parameters of stroke patients initially admitted to a rural primary stroke center (PSC) who receive endovascular treatment (EVT) by a Flying Intervention Team with patients who receive EVT after secondary transfer to a comprehensive stroke center (CSC).

DETAILED DESCRIPTION:
A novel health care concept was implemented in the telemedical stroke network TEMPiS (Telemedical Project for integrative Stroke Care) to reduce time delays to EVT in stroke patients with large vessel occlusion: After telemedicine-assisted identification of EVT candidates in a PSC, a Flying Intervention Team (neuroradiologist and angiography assistant) is flown from a CSC via helicopter to the PSC to perform EVT in the local angiography suite. Flying Intervention Team service runs from 8 a.m. to 10 p.m. Patients remain at local stroke unit for further treatment.

Analysis will include time delay to EVT, recanalization, symptomatic intracerebral hemorrhage, periprocedural complications, in-hospital complications, and mortality.

ELIGIBILITY:
Inclusion criteria:

* Admission to participating primary stroke center (PSC) with acute symptoms of stroke
* Telemedicine-supported decision for endovascular treatment (EVT)

Inclusion criteria for primary study population:

* Occlusion of M1, proximal M2, intracranial internal carotid artery (ICA) or basilar artery
* Decision for EVT between 8 a.m. an 10 p.m.
* Time from symptom onset to EVT decision within treatment window (0-6 h for M1, M2 and ICA occlusions, 0-24 h for basilar artery occlusions, 0-24 for M1, M2 and ICA occlusions with suitable mismatch in perfusion imaging performed in PSC)
* Endovascular treatment in PSC by Flying Intervention Team or in comprehensive stroke center after secondary transfer

Exclusion criteria for primary study population:

* Age > 85 years
* Alberta Stroke Program Early CT score (ASPECTS) < 6
* Premorbid severe or moderately severe disability (modified Rankin Scale > 3)
* Premorbid serious or advanced illness with high mortality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute stroke patients eligible for endovascular treatment initially admitted to participating primary stroke center
Sampling Method: Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Time from decision for endovascular treatment to groin puncture | day 1
  Time from telemedicine-assisted decision for endovascular treatment to initiation of endovascular treatment by groin puncture

SECONDARY OUTCOMES:
Time from symptom onset to recanalization | day 1
  Time from symptom onset to recanalization of previously occluded target artery by endovascular treatment
Other procedural times of hyperacute care | day 1
  Other procedural times between symptom onset, admission to PSC, first imaging, decision for endovascular treatment, initiation of endovascular treatment and completion of endovascular treatment
Recanalization | day 1
  Proportion of patients with antegrade reperfusion of more than half of the previously occluded target artery ischemic territory after endovascular treatment
Symptomatic intracerebral hemorrhage | 7 days
  Proportion of patients with symptomatic intracerebral hemorrhage
In-hospital death or palliative care | 7 days
  In-hospital death or decision for palliative care
Periprocedural complications | day 1
  Proportion of patients with periprocedural, endovascular treatment associated complications
In-hospital complications | 7 days
  Proportion of patients with other in-hospital complications

CONTACTS AND LOCATIONS:
Overall Officials: Gordian J Hubert, Dr. med., Principal Investigator — München Klinik gGmbH
Locations (1):
- TEMPiS TeleStroke Network, Department of Neurology, Munich Municipal Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Saver JL, Goyal M, van der Lugt A, Menon BK, Majoie CB, Dippel DW, Campbell BC, Nogueira RG, Demchuk AM, Tomasello A, Cardona P, Devlin TG, Frei DF, du Mesnil de Rochemont R, Berkhemer OA, Jovin TG, Siddiqui AH, van Zwam WH, Davis SM, Castano C, Sapkota BL, Fransen PS, Molina C, van Oostenbrugge RJ, Chamorro A, Lingsma H, Silver FL, Donnan GA, Shuaib A, Brown S, Stouch B, Mitchell PJ, Davalos A, Roos YB, Hill MD; HERMES Collaborators. Time to Treatment With Endovascular Thrombectomy and Outcomes From Ischemic Stroke: A Meta-analysis. JAMA. 2016 Sep 27;316(12):1279-88. doi: 10.1001/jama.2016.13647. PMID 27673305
- [Background] Jahan R, Saver JL, Schwamm LH, Fonarow GC, Liang L, Matsouaka RA, Xian Y, Holmes DN, Peterson ED, Yavagal D, Smith EE. Association Between Time to Treatment With Endovascular Reperfusion Therapy and Outcomes in Patients With Acute Ischemic Stroke Treated in Clinical Practice. JAMA. 2019 Jul 16;322(3):252-263. doi: 10.1001/jama.2019.8286. PMID 31310296
- [Derived] Leitner MA, Hubert GJ, Paternoster L, Leitner MI, Remi JM, Trumm C, Haberl RL, Hubert ND. Clinical outcome of rural in-hospital-stroke patients after interhospital transfer for endovascular therapy within a telemedical stroke network in Germany: a registry-based observational study. BMJ Open. 2024 Jan 18;14(1):e071975. doi: 10.1136/bmjopen-2023-071975. PMID 38238050
- [Derived] Hubert GJ, Kraus F, Maegerlein C, Platen S, Friedrich B, Kain HU, Witton-Davies T, Hubert ND, Zimmer C, Bath PM, Audebert HJ, Haberl RL. The "Flying Intervention Team": A Novel Stroke Care Concept for Rural Areas. Cerebrovasc Dis. 2021;50(4):375-382. doi: 10.1159/000514845. Epub 2021 Apr 13. PMID 33849042
- See also: TEMPIS — http://www.tempis.de/